CLINICAL TRIAL: NCT03320434
Title: A Single-Center, Randomized, Double-Masked, Vehicle and Active-Controlled, Dose-Ranging Phase 2 Study Evaluating the Efficacy and Safety of PRT-2761 for the Treatment of Acute and Chronic Allergic Conjunctivitis Using the Conjunctival Allergen Challenge Model (Ora-CAC®)
Brief Title: Study Evaluating the Efficacy and Safety of PRT-2761 for the Treatment of Acute and Chronic Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-100-0008
Record Dates: First submitted 2017-10-19; First posted 2017-10-25 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PRT-2761 0.5% (Experimental)
  Interventions: Drug: PRT-2761 0.5%
- PRT-2761 1% (Experimental)
  Interventions: Drug: PRT-2761 1%
- Patanol (Active Comparator)
  Interventions: Drug: Patanol
- Pred-forte (Active Comparator)
  Interventions: Drug: Pred-forte
- PRT-2761 0% (Placebo Comparator)
  Interventions: Drug: PRT-2761 0%

INTERVENTIONS:
Drug: PRT-2761 0.5% — Six drops in each eye over a 17 day period.
  Arms: PRT-2761 0.5%
Drug: PRT-2761 1% — Six drops in each eye over a 17 day period.
  Arms: PRT-2761 1%
Drug: Patanol — Six drops in each eye over a 17 day period.
  Arms: Patanol
Drug: Pred-forte — Four drops in each eye over a 3 day period.
  Arms: Pred-forte
Drug: PRT-2761 0% — Six drops in each eye over a 17 day period.
  Arms: PRT-2761 0%

SUMMARY:
To evaluate the efficacy and safety of two concentrations of PRT-2761 as a topical ophthalmic solution for the treatment of the signs and symptoms of acute and chronic allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years old
* be willing and able to avoid all disallowed medications and contact lenses
* must have a pregnancy test if of childbearing potential
* must be able to read an eye chart from 10 feet away

Exclusion Criteria:

* must not have any allergies to the study medications
* must not have any ocular or non ocular condition that investigator feels will interfere with study parameters
* must not have used an investigational drug or device in the past 30 days or concurrently enrolled in another investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one site in the US.
Pre-assignment Details: One hundred and twenty participants enrolled and 97 subjects completed the study. Participant flow and baseline characteristics are presented for 120 subjects that met all inclusion, none of the exclusion criteria, and were randomized to receive one of five treatments based on the randomization list.
Period: Overall Study
Arm/Group | PRT-2761 0.5% | PRT-2761 1% | Patanol | PRT-2761 0%
Started | 32 | 29 | 30 | 29
Completed | 25 | 23 | 28 | 23
Not Completed | 7 | 6 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRT-2761 0.5% | PRT-2761 1% | Patanol | PRT-2761 0% | Total
Number analyzed (Participants) | 32 | 29 | 30 | 29 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 27 | 30 | 27 | 114
  >=65 years | 2 | 2 | 0 | 2 | 6
Age, Continuous [Median (Standard Deviation); unit: years] | 52 (14.49) | 49 (12.98) | 46 (10.81) | 52 (9.21) | 50 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 16 | 15 | 67
  Male | 8 | 17 | 14 | 14 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 3 | 5 | 20
  Not Hispanic or Latino | 29 | 20 | 27 | 24 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 0 | 2 | 4 | 9
  White | 29 | 27 | 27 | 23 | 106
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 29 | 30 | 29 | 120
Iris Color [Count of Participants; unit: Participants]
  Black | 0 | 0 | 0 | 2 | 2
  Blue | 10 | 12 | 8 | 6 | 36
  Brown | 13 | 12 | 15 | 17 | 57
  Hazel | 4 | 4 | 5 | 1 | 14
  Green | 5 | 1 | 2 | 3 | 11
Average Post-CAC Itching Score at Baseline [Count of Participants; unit: Participants]
  ≤ 2.5 | 7 | 5 | 6 | 5 | 23
  > 2.5 | 25 | 24 | 24 | 24 | 97
Allergen Type [Count of Participants; unit: Participants]
  Seasonal | 22 | 21 | 20 | 20 | 83
  Perennial | 10 | 8 | 10 | 9 | 37
Confocal Participation [Count of Participants; unit: Participants]
  Yes | 11 | 8 | 10 | 8 | 37
  No | 21 | 21 | 20 | 21 | 83

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching at 5, 7, and 10 Minutes Post CAC on Day 1
Description: Ocular Itching was assessed by a trained investigator post-conjunctival allergen challenge (CAC) on a 0 to 4 scale (0=none (best/no itching) to 4=severe (worst/most itching). The ocular itching was averaged across all subjects at each time point.
Time Frame: post CAC exposure at 5, 7, and 10 minutes post CAC on Day 1
Population: All Randomized Participants Population - All participants who received study treatment.
  Note: Pred forte subjects receive Patanol up to and including Visit 5a and are analyzed as Patanol subjects for those visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRT-2761 0.5% | PRT-2761 1% | Patanol | PRT-2761 0%
Number analyzed (Participants) | 32 | 29 | 30 | 29
units on a scale
  5 minutes post-CAC: number analyzed (Participants) | 31 | 29 | 30 | 29
  5 minutes post-CAC | 2.573 (0.9246) | 2.500 (0.7792) | 1.217 (0.8826) | 2.647 (0.8170)
  7 minutes post-CAC: number analyzed (Participants) | 31 | 29 | 30 | 29
  7 minutes post-CAC | 2.677 (0.8879) | 2.509 (0.8114) | 1.358 (0.8627) | 2.629 (0.7459)
  10 minutes post-CAC: number analyzed (Participants) | 31 | 29 | 30 | 29
  10 minutes post-CAC | 2.250 (1.0878) | 2.293 (1.0135) | 1.258 (0.9727) | 2.190 (0.8754)

2. Primary Outcome: Ocular Itching at 5, 7, and 10 Minutes Post CAC on Day 15
Description: Ocular Itching was assessed by the subjects using a 0 to 4 point scale(0=none (best/no itching) to 4=severe (worst/most itching)). The ocular itching was averaged across all subjects at each time point.
Time Frame: post CAC exposure at 5, 7, and 10 minutes post CAC on Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRT-2761 0.5% | PRT-2761 1% | Patanol | PRT-2761 0%
Number analyzed (Participants) | 32 | 29 | 30 | 29
units on a scale
  5 minutes post-CAC: number analyzed (Participants) | 29 | 27 | 30 | 28
  5 minutes post-CAC | 2.431 (1.1415) | 2.611 (0.7731) | 0.775 (0.7172) | 2.527 (0.9288)
  7 minutes post-CAC | 2.362 (1.0724) | 2.602 (0.7883) | 0.808 (0.7505) | 2.366 (0.9317)
  10 minutes post-CAC: number analyzed (Participants) | 29 | 27 | 30 | 28
  10 minutes post-CAC | 1.922 (1.1242) | 2.204 (1.0630) | 0.833 (0.8077) | 1.929 (0.9425)

3. Primary Outcome: Conjunctival Redness at 7, 15, and 20 Minutes Post CAC on Day 1
Description: Conjunctival Redness was assessed by a trained investigator post-conjunctival allergen challenge (CAC) on a 0 to 4 scale (0=none (best/no redness) to 4=severe (worst/most redness)).
  The conjunctival redness was averaged across all subjects at each time point.
Time Frame: post CAC exposure at 7, 15, and 20 minutes post-CAC on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRT-2761 0.5% | PRT-2761 1% | Patanol | PRT-2761 0%
Number analyzed (Participants) | 32 | 29 | 30 | 29
units on a scale
  7 minutes post-CAC: number analyzed (Participants) | 31 | 29 | 30 | 29
  7 minutes post-CAC | 1.282 (0.6479) | 1.491 (0.5919) | 1.592 (0.7236) | 1.957 (0.4913)
  15 minutes post-CAC: number analyzed (Participants) | 31 | 29 | 30 | 29
  15 minutes post-CAC | 1.411 (0.6142) | 1.526 (0.5989) | 1.833 (0.7350) | 2.181 (0.3774)
  20 minutes post-CAC: number analyzed (Participants) | 31 | 29 | 30 | 29
  20 minutes post-CAC | 1.371 (0.5841) | 1.603 (0.6251) | 1.917 (0.6833) | 2.164 (0.4496)

4. Primary Outcome: Conjunctival Redness at 7, 15, and 20 Minutes Post CAC on Day 15
Description: as for outcome 3
Time Frame: post CAC exposure at 7, 15, and 20 minutes post-CAC on Day 15.
Population: All Randomized Participants Population - All participants who received study treatment.
  Note: Pred forte subjects receive Patanol up to and including Visit 5a.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRT-2761 0.5% | PRT-2761 1% | Patanol | PRT-2761 0%
Number analyzed (Participants) | 32 | 29 | 30 | 29
units on a scale
  7 minutes post-CAC: number analyzed (Participants) | 28 | 27 | 30 | 28
  7 minutes post-CAC | 1.723 (0.5787) | 2.056 (0.4458) | 1.242 (0.7296) | 1.973 (0.4731)
  15 minutes post-CAC: number analyzed (Participants) | 28 | 27 | 30 | 28
  15 minutes post-CAC | 1.920 (0.6703) | 2.176 (0.4894) | 1.617 (0.7478) | 1.991 (0.5464)
  20 minutes post-CAC: number analyzed (Participants) | 28 | 27 | 30 | 28
  20 minutes post-CAC | 1.857 (0.6289) | 2.222 (0.6699) | 1.592 (0.7266) | 2.036 (0.6372)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 9 weeks. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited, or observed.
Arm/Group | PRT-2761 0.5% | PRT-2761 1% | Patanol | PRT-2761 0%
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 4/32 | 9/29 | 1/30 | 7/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRT-2761 0.5% (N=32) | PRT-2761 1% (N=29) | Patanol (N=30) | PRT-2761 0% (N=29)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival Pigmentation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal Opacity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid Oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meibomian Gland Dysfunction (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Punctate Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT03320434/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03320434/SAP_001.pdf